CLINICAL TRIAL: NCT05396183
Title: A Prospective Single-arm Cohort Study on Accuracy and Safety of Coplanar Template Assisted CT-guided Neck and Head Biopsies.
Brief Title: Accuracy and Safety of Coplanar Template Assistance for Head and Neck Biopsies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Peking University, Peking University Third Hospital
Other Study IDs: ChiECRCT20220052
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms; biopsy; 3D-PCT
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D-PCT group: Participant will receive three-dimensional printing co-planar template (3D-PCT) assisted CT-guided head and neck neoplasm biopsy and prospective accuracy and safety data will record.

SUMMARY:
This is a prospective single-arm cohort study to evaluate the accuracy and safety of three-dimensional printing co-planer template(3D-PCT) for computed tomography (CT)-guided neck and head biopsy .

DETAILED DESCRIPTION:
Tumors in head and neck region refer to those located above the clavicle, the upper boundary is the skull base, the posterior boundary is cervical vertebra, excluding brain spinal cord and other central nervous system and Intraocular tumor. Include oral cavity (lips, tongue, hard palate, floor of mouth, gums), oropharynx (middle of throat behind mouth, including tongue base, tonsils, and soft palate), larynx, hypopharynx (lower throat), paranasal sinuses, nasopharynx, salivary glands (Parotid, submandibular and minor salivary glands), thyroid, skin cancers and metastatic cancers of the head and neck. Tissue sampling of lesions in the head and neck is limited due to the complex regional anatomy, including nerves, vessels, and salivary glands. Computed tomography (CT)-guided percutaneous puncture biopsy is a well-recognized technique that can facilitate histopathological diagnosis and therapeutic planning of head and neck masses, and may be particularly useful when lesions are not accessible via an endoscope or by palpation-guided sampling. CT image-guided free-hand puncture biopsy is widely used in clinical practice. However, multiple CT scan and adjustment of position of the biopsy needle increased radiation exposure and the probability of other adverse events, such as bleeding and nerve injury. Therefore, we need a more efficient approach to guidance which is precisely positioned and safe to operate.

In recent years, we have taken advantage of three-dimensional(3D) printing template to improve the accuracy and safety of puncture related operations, which simplifies the procedure and shortens the procedure duration[3-4]. 3D printing template include co-planar and non co-planar[5]. However, few prospective studies have focused on three-dimensional printing co-planer template(3D-PCT) for CT-guided neck and head biopsy. The purposes of this prospective, single-arm study are to determine the accuracy and safety of CT guided percutaneous head and neck biopsy assisted by 3D-PCT.

1. Tu A S, Geyer C A, Mancall A C, et al. The buccal space: A doorway for percutaneous CT-guided biopsy of the parapharyngeal region. Am J Neuroradiol, 1998.19（4）：728- 731.
2. Esposito M B, Arrington J A, Murtagh F R, et al. Anterior approach for CT-guided biopsy of skull base and parapharyngeal space lesions. J Comput Assist Tomogr, 1996. 20 (5)：739-741.
3. Ji Z, Jiang Y ,Guo F, et al. Dosimetry verification of radioactive seed implantation for malignant tumor assisted by 3D printing individual templates and CT guidance. Applied Radiation and lsotopes 2017; 124: 68-74.
4. Jiang Y, Ji Z , Guo F, et al. Side effects of CT-guided implantation of 125I seeds for recurrent malignant tumors of the head and neck assisted by 3D printing non co-planar template[J]. Radiation Oncology, 2018, 13(1):18.
5. W J, Chai S, Wang R, et al. Expert consensus on computed tomography-assisted three-dimensional-printed coplanar template guidance for interstitial permanent radioactive (125) I seed implantation therapy. J Cancer Res Ther 2019; 15: 1430-1434.

ELIGIBILITY:
Inclusion Criteria:

(1) Ages 18 to 80; (2) KPS>70 points, an estimated life expectancy of greater than 3 months; (3)Head and neck masses or nodules can be revealed by CT scan, MRI or ultrasonic examination; (4) Without taking drugs affecting coagulation and/or platelet aggregation are used; If used, the drug has been discontinued for a sufficient period of time (e.g. 1 week) ; (5) No serious or uncontrolled underlying diseases, clinical evaluation patients can tolerate puncture; (6) Planned biopsy with applicable puncture path; (7) With informed consent.

Exclusion Criteria:

(1)Biopsy needle insertion route impeded by skeletal structures and close to blood vessels which have high risks of puncture bleeding; (2)Poor organ function (e.g. poorly controlled high blood pressure); (3) Any contraindication of percutaneous head and neck biopsy; (4) Poor compliance, unable to complete coordination; (5) Participant who is considered inappropriate or unwilling to participate in this clinical trial for other reasons.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible patient with head and neck masses or nodules, who are planned undergo biopsy with applicable puncture path in Peking university Third hospital will be enrolled.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
Accuracy | During the operation.
  Depth and Angle difference between actual puncture and planned puncture pathway.

SECONDARY OUTCOMES:
Complication rate | During the first month after operation.
  Adverse event include needle track implantation metastasis and operation-related complications (e.g. bleeding, nerve injury, air embolism).
Pathological Diagnosis | During the first month after operation.
  The pathological diagnosis of head and neck biopsy.

OTHER OUTCOMES:
Procedural duration | During the operation.
  The length of procedural duration was measured from the time a patient lain on the examining bed of the CT scanner to the time the first CT scan post biopsy.
Radiation exposure | During the operation.
  Numbers of CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Junjie, Principal Investigator — Peking University Third Hospital
Locations (1):
- Department of Radiation Oncology of Peking university third hospital, Beijing, Beijing Municipality, China